CLINICAL TRIAL: NCT03442855
Title: Non-Interventional, Multicenter Bicontact® E PMCF Study
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1417
Record Dates: First submitted 2018-02-06; First posted 2018-02-22 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Degenerative Osteoarthritis; Rheumatoid Arthritis; Femoral Neck Fractures; Femoral Head Necrosis
Keywords: Arthroplasty, Replacement, Hip
MeSH Terms: conditions — Joint Diseases; Arthritis, Rheumatoid; Femoral Neck Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective observational (non-interventional) cohort study, multi-centric in 5 study Centers in Japan to collect short term clinical and radiological results of the cementless Bicontact® E stem in a standard patient population used in routine clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Indication for Bicontact E prosthesis THA
* Patients ≥ 18 years
* Patient not pregnant
* Written informed consent

Exclusion Criteria:

- Patients receiving a bipolar implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving primary THA:
  Acute disorders of the hip that cannot be treated by other therapies:
  * Degenerative osteoarthritis
  * Rheumatic arthritis
  * Joint fractures
  * Femoral head necrosis
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Clinical Results | 1 year
  Hip Score of the Japanese Orthopaedic Association (JOA): three categories-movement, mental, and pain-each comprising 7 items, for a total of 21 items to be used as evaluation criteria for hip-joint function

SECONDARY OUTCOMES:
Thigh Pain | 1 year
  Pain as measured with the Visual Analog Scale (VAS): Visual analog scale [VAS] is a measure of pain intensity. It is a continuous scale comprised of a horizontal analog scale of 100 mm length. It is anchored by two verbal descriptors, one for each symptom extreme [no pain - worst imaginable pain].
X-Ray evaluation | 1 year
  Radiological results (osteointegration, migration)
(Serious) Adverse Events | 1 year
  Complications: Adverse Events (AE) / Serious Adverse Events (SAE)

CONTACTS AND LOCATIONS:
Locations (5):
- Japan (5):
  - Funabashi Orthopedic Hospital, Funabashi
  - Niigata Bandai Hospital, Niigata
  - Niigata Rinko Hospital, Niigata
  - Niigata Univ. Medical & Dental Hospital, Niigata
  - Saiseikai Niigata Second Hospital, Niigata